CLINICAL TRIAL: NCT04505566
Title: INflammatory MediatorS in the PathophysIology of Diabetic REtinopathy (INSPIRE) Study
Brief Title: INflammatory MediatorS in the PathophysIology of Diabetic REtinopathy Study
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stephen J. Kim, MD (Other)
Collaborators: Allergan (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Stephen J. Kim, MD, Professor of Ophthalmology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201433; 5R01EY031315-02 (NIH)
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Retinopathy
Keywords: Topical Ketorolac; Acuvail; Prevention of Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ketorolac; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This is a 2 aim, randomized and double-masked Phase I study on topical Ketorolac for the prevention of diabetic retinopathy.
  164 adult type II diabetic patients, aged 18 years or greater will be enrolled in addition to 100 age-matched patients without diabetes who are undergoing unilateral vitrectomy surgery for non-inflammatory conditions such as epiretinal membrane or macular hole will also be enrolled.
Who Masked: Participant, Investigator
Masking Description: At the baseline visit, only patients from the moderate NPDR group will be randomized into one of 2 groups, using a red cap database for randomization in a block manner to ensure near equal randomization in both groups.
  A report is generated every 4 months for assessment of the number of patients in each randomized category.
  Patients in this group will have both eyes randomized to either Acuvail or placebo-control (preservative-free artificial tear) in double-masked fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Adult Type II Diabetics - Moderate NPDR - Ketorolac (Experimental): 59 Adult type II diabetic patients with baseline moderate non-proliferative diabetic retinopathy and HbA1c ≥ 8 randomized to Ketorolac treatment.
  Interventions: Drug: Ketorolac 0.45% ophthalmic solution; Other: Aqueous PGE2 and inflammatory cytokines measurements
- Adult Type II Diabetics - Moderate NPDR - Placebo (Placebo Comparator): 59 Adult type II diabetic patients with baseline moderate non-proliferative diabetic retinopathy randomized to placebo treatment.
  Interventions: Drug: Placebo - Preservative-free artificial tears; Other: Aqueous PGE2 and inflammatory cytokines measurements
- Adult Type II Diabetics - No Diabetic Retinopathy (DR) (Other): 23 Adult type II diabetic patients with no diabetic retinopathy as a control group.
  Interventions: Other: Aqueous PGE2 and inflammatory cytokines measurements
- Adult Type 2 Diabetics-Proliferative Diabetic Retinopathy(PDR) (Other): 23 Adult type II diabetic patients with proliferative diabetic retinopathy as a control group.
  Interventions: Other: Aqueous PGE2 and inflammatory cytokines measurements
- Age-matched Non-diabetics (Other): We will also enroll 100 age-matched patients without diabetes who are undergoing unilateral vitrectomy surgery for non-inflammatory conditions such as epiretinal membrane or macular hole. Removed aqueous fluid that is typically discarded will instead be collected and stored at -80° C. Aqueous fluid will be tested for inflammatory markers as detailed below to provide a reference level for cross-comparison analysis.
  Interventions: Other: Aqueous PGE2 and inflammatory cytokines measurements

INTERVENTIONS:
Drug: Ketorolac 0.45% ophthalmic solution — Ketorolac 0.45% ophthalmic solution 1 drop instilled in both eyes twice daily for 3 years in double-masked fashion.
  Other Names: Acuvail
  Arms: Adult Type II Diabetics - Moderate NPDR - Ketorolac
Drug: Placebo - Preservative-free artificial tears — Preservative free artificial tears ophthalmic solution 1 drop instilled in both eyes twice daily for 3 years in double-masked fashion.
  Other Names: Refresh
  Arms: Adult Type II Diabetics - Moderate NPDR - Placebo
Other: Aqueous PGE2 and inflammatory cytokines measurements — After topical anesthetic, antibiotic and 5% povidone-iodine application, a 30 gauge needle on a 1 ml tuberculin syringe will be inserted into the anterior chamber and used to collect 0.1 ml of aqueous fluid from each eye. Aqueous PGE2 and Inflammatory cytokines will be measured

SUMMARY:
The central hypothesis is that inflammation mediators are biomarkers of both systemic diabetes and Diabetic Retinopathy (DR) progression in the aqueous and that sustained topical ketorolac application reduces/suppresses those inflammatory mediators thereby reducing the progression of Diabetic Retinopathy.

DETAILED DESCRIPTION:
Study goals include confirming inflammation mediators are biomarkers of both systemic diabetes and DR progression in the aqueous. Like the vitreous humor, the aqueous reflects localized ocular inflammation, however, is technically easier to collect with less risk. The investigators will also determine the long-term effects of sustained ketorolac application on intraocular cytokine levels, DR progression, and diabetic macular edema (DME) incidence. The proposal is the first to use a cornea-permeable Nonsteroidal anti-inflammatory drug (NSAID) for the treatment of DR.

It is believed local inflammation control in the eye will transform future treatment options for diabetic patients facing blindness. Tracking and inhibiting local inflammatory mediators through all DR stages has the capacity to reduce or prevent disability in millions of patients per year.

164 adult type II diabetic mellitus (T2DM) patients, aged 18 years or greater will be enrolled to measure aqueous PGE2 and inflammatory cytokines. Because the pathophysiology of type I disease and the population it effects are different, type I diabetic patients will be excluded. Diabetic retinopathy is broadly categorized as nonproliferative (NPDR) and proliferative (PDR). The international Clinical Disease Severity Scale is a standard classification system consisting of two categories and five stages: the nonproliferative category, stage 1-4 and proliferative category, stage 5. Stage 1 is characterized as "no apparent retinopathy." The nonproliferative stage is further grouped into stage 2 (mild), stage 3 (moderate), and stage 4 (severe). Stage 5 is final stage, PDR.

Of the 164 patients enrolled for aqueous PGE2 and inflammatory cytokine measurements, the diabetic participants corresponding to stages 1, 3, and 5 will be classified as patients with no DR (23 patients), with PDR (23 patients), and with moderate NPDR (118 patients). The 118 participants with moderate NPDR will be randomized for Aim 2 described below.

In addition, 100 age-matched patients without diabetes who are undergoing unilateral vitrectomy surgery for non-inflammatory conditions such as epiretinal membrane or macular hole will be enrolled as controls.

Aim 1 of this project is to measure aqueous PGE2 and inflammatory cytokines during DR progression.

Aim 2 of this project is two-fold:

1. Investigate the long-term effects of daily topical application of ketorolac on PGE2 and cytokine levels.
2. Determine how topical application of ketorolac influences DR progression and development of DME.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1 Diabetic Arm Inclusion Criteria: Adult patients age 18 years or greater with type II diabetes.
* Aim 1 Nondiabetic Control Arm Inclusion Criteria: age-matched patients without diabetes who are undergoing unilateral vitrectomy surgery for non-inflammatory conditions such as epiretinal membrane or macular hole.
* Aim 2 Inclusion Criteria: Adult patients age 18 years or older with type II diabetes, with baseline moderate NPDR and HbA1c ≥ 8.

Exclusion Criteria:

* Aim 1 Diabetic Arm Exclusion Criteria: Patients with a history of previous vitrectomy in either eye; prior intravitreal injection within 3 months; co-existent macular, retinovascular, or inflammatory disease; history of ocular trauma; aphakia; presence of an anterior chamber intraocular lens; current use of prescription systemic NSAIDs or regular use of nonprescription NSAIDs including aspirin (defined as 4 days or more a week for at least 2 weeks a month); blood pressure > 180/110 mmHg; risk for corneal melting; and inability to comply with follow-up.
* Aim 1 Nondiabetic Control Arm Exclusion Criteria: Patients who are unable to comply with testing and follow-up.
* Aim 2 Exclusion Criteria: Patients with a history of previous vitrectomy in either eye; prior intravitreal injection within 3 months; co-existent macular, retinovascular, or inflammatory disease; history of ocular trauma; aphakia; presence of an anterior chamber intraocular lens; current use of prescription systemic NSAIDs or regular use of nonprescription NSAIDs including aspirin (defined as 4 days or more a week for at least 2 weeks a month); blood pressure > 180/110 mmHg; risk for corneal melting; and inability to comply with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PGE2 level during Diabetic Retinopathy progression | 1 year
  Aqueous samples will be analyzed using liquid chromatography electrospray ionization tandem mass spectrometry to measure all PGE2 levels. PGE2 will be measured every 4 months during 1 year of study to determine whether their mean mediator levels associate with DR severity stage using a linear mixed effects model. The DR severity stage will be included as a continuous or categorical variable, and potential confounding factors as well as baseline measurements for each inflammatory mediator, will be adjusted in the analysis.
Vascular Endothelial Growth Factor (VEGF) level during Diabetic Retinopathy progression | 1 year
  Aqueous samples will be analyzed using a microparticle bead-based multiplex assay will be used to measure VEGF levels. VEGF will be measured every 4 months during 1 year of study to determine whether their mean mediator levels associate with DR severity stage using a linear mixed effects model. The DR severity stage will be included as a continuous or categorical variable, and potential confounding factors as well as baseline measurements for each inflammatory mediator, will be adjusted in the analysis.
Interleukin 6 (IL-6) level during Diabetic Retinopathy progression | 1 year
  Aqueous samples will be analyzed using a microparticle bead-based multiplex assay will be used to measure IL-6 levels. VEGF will be measured every 4 months during 1 year of study to determine whether their mean mediator levels associate with DR severity stage using a linear mixed effects model. The DR severity stage will be included as a continuous or categorical variable, and potential confounding factors as well as baseline measurements for each inflammatory mediator, will be adjusted in the analysis.
Interleukin 8 (IL-8) level during Diabetic Retinopathy progression | 1 year
  Aqueous samples will be analyzed using a microparticle bead-based multiplex assay will be used to measure IL-8 levels. VEGF will be measured every 4 months during 1 year of study to determine whether their mean mediator levels associate with DR severity stage using a linear mixed effects model. The DR severity stage will be included as a continuous or categorical variable, and potential confounding factors as well as baseline measurements for each inflammatory mediator, will be adjusted in the analysis.
Progression of Diabetic Retinopathy (DR) | 3 years
  To determine progression of DR, we will analyze data from the 118 diabetic patients randomized to either Ketorolac or placebo. Diabetic retinopathy progresses in discrete steps defined by the Early Treatment Diabetic Retinopathy Study (ETDRS) severity scale (15-step scale: minimum value of 10 and maximum value of 65, with higher scores meaning a worse outcome). With each advancing level, the risk of developing DME and/or PDR increases. A 2-stage or more worsening on the ETDRS severity scale is associated with an increased risk of vision loss.
Severity of Diabetic Retinopathy (DR) | 3 years
  A blinded sub-investigator will grade DR by utilizing the 15-step severity scale established by the ETDRS. A 2-step or more increase or decrease in severity scale, observed on 2 consecutive follow-up appointments, will define a change in DR (progression or improvement).

SECONDARY OUTCOMES:
Incidence of Diabetic Macular Edema | 3 years
  To determine incidence of Diabetic Macular Edema, we will analyze data from the 118 diabetic patients. An increase in macular thickness (determined by OCT as ≥ 40%) will determine development of DME.
Progression of Diabetic Macular Edema | 3 years
  To determine progression of Diabetic Macular Edema, we will analyze data from the 118 diabetic patients. An increase in macular thickness (determined by OCT as ≥ 40%) will determine progression of DME.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Kim SJ, Gangaputra S, Sheng J, Patel S, Nair AA, Al Hussein Al Awamlh S, Fitzpatrick J, Cherney E, Veach L, Nicholson C. Analysis of 24 pro-inflammatory cytokines in aqueous and serum of 94 patients without diabetes. Br J Ophthalmol. 2025 Nov 20;109(12):1357-1362. doi: 10.1136/bjo-2025-327421. PMID 40695570